CLINICAL TRIAL: NCT06984185
Title: Contribution of a Combined T1D Autoantibody Test and Immunoreactive Trypsin Assay on Blotting Paper in the Detection of Type 1 Diabetes (Stage 3) in the Pediatric Population With a View to Its Subsequent Use in Early Detection (Stages 1 and 2)
Brief Title: Early Detection of Type 1 Diabetes
Acronym: PREDIDIA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_1022
Record Dates: First submitted 2025-04-28; First posted 2025-05-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; children; prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anti-GAD, anti-IA2 and anti-ZNT8 antibodies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PREDIDIA: Pediatric patients (1-18 years) with suspicion of type 1 diabetes at stage 3
  Interventions: Diagnostic Test: combined assay on capillary blotting paper

INTERVENTIONS:
Diagnostic Test: combined assay on capillary blotting paper — combined assay on capillary blotting paper

SUMMARY:
T1D is an autoimmune disease characterized by the presence of autoantibodies usually assayed separately on venous blood. The use of a combined test on capillary blood using a blotting paper would facilitate the immunological presymptomatic T1D screening in routine clinical practice as it is easy to perform and can be performed at home by families.

However the use of a combined test on blotting paper must be validated before it is used in routine clinical practice for preclinical T1D screening purpose at large scale, starting with pediatric first degree relatives of T1D patients: this is the aim of this study, where we will assess the concordance of 3 autoantibodies rates (anti-GAD65, anti-IA2 and anti-ZnT8) between a combined assay on capillary blotting paper and the individual measurement of these 3 autoantibodies in venous blood at the time of discovery of type 1 diabetes (stage 3).

The combined immunological test used in this study has already been validated (test available on the market: (Biosynex - product code: RL 3ZGl/96D); However, it has never been used on capillary blood eluate from blotting paper. The blotting paper to be used is also marketed and used in current clinical practice for newborn screening (test WHATMAN® + SAVER CARDS 903x100 - ref: 034955).

Of note: this ELISA 3 screen test does not include IAA. In clinical practice, for stage 3 patients, IAA (from venous samples) is systematically tested for children < 6-year-old. For older children they are tested only if the other 3 autoantibodies are negative. (IAA are found more commonly in young children and mainly below 4 years old and mark a higher risk of progression at a very young age. A single IAA positivity in children can therefore justify a closer surveillance in the short term).

HCL choose to validate the combined assay (3 Screen + blotting paper) in symptomatic children with suspicion of type 1 diabetes at stage 3, to be further used for pre-clinical T1D screening activities across Auvergne Rhone-Alpes region.

3-screen tests have already been used in large screening program (FR1DA). Added to this, any positivity must be confirmed by a second measurement of all 4 individual Aabs on a venous blood sample within 3 months of the positive screening according to the French recommendation.

In addition, although it is usual to consider that the attack is targeted in the islets of Langerhans with the destruction of beta cells, the exocrine pancreas is also the site of inflammation, leading to the rapid reduction of the mass of the pancreas, which can impact beta cell function and accelerate the autoimmune process of T1D. With this regard, the level of immunoreactive trypsin on blotting paper could be an early marker of the progression of T1D.

The secondary objective of the study is therefore to verify if levels of immunoreactive trypsin on blotting paper, at the time of discovery of type 1 diabetes (stage 3) in pediatric age, is decreased compared to general pediatric population levels. Trypsin measurements will be performed in the study from the same blotting paper and veinous sample as for Aabs. They will be compared to normal values from general population on venous blood and blotting paper (neonatal screening). If trypsin levels are collapsed in stage 3, this marker could be studied in early stages of diabetes and could be an early marker of progression to stage 3, then useful for monitoring early stages. Further studies would then be necessary.

Overview/Hypothesis:

The research hypothesis are that i) the combined assay of anti-GAD65, anti-IA2 and anti-ZnT8 autoantibodies by a combined capillary blotting paper test is equivalent to the individual measurement of these 3 autoantibodies on venous sampling at the time of discovery of stage 3 type 1 diabetes and ii) capillary levels of immunoreactive trypsin on blotting paper, at the time of discovery of type 1 diabetes (stage 3) in pediatric age, is decreased compared to normal values (in general pediatric population) and could be a prognostic marker.

ELIGIBILITY:
Inclusion criteria:

* Children aged over 1 year and under 18 years
* BMI <30.0 kg/m2
* With a diagnosis of stage 3 type 1 diabetes (clinical and laboratory criteria, metabolic acidosis, ketone levels)
* Child's consent and no parental opposition Exclusion criteria
* Patients with T2D or monogenic diabetes with a known familial history
* Patients with cystic fibrosis
* History of liver or kidney disease, or pancreatitis
* Any progressive disease (other than T2D)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (1-18 years) with suspicion of type 1 diabetes at stage 3
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Concordance rate between the autoantibodies combined assay and the individual assays | Day 1
  To assess the concordance of the 3 autoantibodies rates (anti-GAD65, anti-IA2 and anti-ZnT8) between a combined assay on capillary blotting paper and the individual measurement of the 3 autoantibodies in venous blood at the time of discovery of type 1 diabetes (stage 3)

CONTACTS AND LOCATIONS:
Locations (1):
- Femme Mère Enfant Hospital, Hospices Civils de Lyon, Bron, Rhône, France

IPD SHARING:
Plan to Share IPD: No